CLINICAL TRIAL: NCT04171570
Title: DISCO Radial Trial: DIStal Versus COnventional RADIAL Access for Coronary Angiography and Intervention: a Randomized Multicenter Trial
Brief Title: DIStal Versus COnventional RADIAL Access for Coronary Angiography and Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: T133E3
Record Dates: First submitted 2019-10-23; First posted 2019-11-21 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Coronary Disease
Keywords: Distal Transradial Access; Randomized Multicenter Trial; Radial Access
MeSH Terms: conditions — Coronary Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Randomization to distal transradial access or conventional transradial access. Both techniques are standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal Transradial Access (Other): Distal Transradial Access
  Interventions: Procedure: Coronary angiography and or Percutaneous coronary Intervention
- Conventional Transradial Access (Other): Conventional Transradial Access
  Interventions: Procedure: Coronary angiography and or Percutaneous coronary Intervention

INTERVENTIONS:
Procedure: Coronary angiography and or Percutaneous coronary Intervention — Radial access punture site

SUMMARY:
The objective of this study is to demonstrate the superiority of Distal Radial Access (DTRA) to Conventional Transradial Access (CTRA) regarding forearm radial artery occlusion (RAO).

This trial plans to include 1300 patients in around 12 locations around the world (11 participating sites in Europe and 1 participating site in Japan).

DETAILED DESCRIPTION:
DISCO RADIAL is a prospective, global, open label, multi-centre randomized controlled trial with plan to include approximately 1300 patients on who transradial coronary angiography and/or intervention is performed. The patients will be randomized in 1:1 ratio to either Distal Transradial Artery Access (DTRA) or Conventional Transradial Access (CTRA) arm. In both arms 6Fr Glidesheath Slender (GSS) will be used as access sheath.

The sponsor will work in accordance with standard operating procedures (SOP) and the Monitoring Plan in order to ensure adherence to the CIP and applicable regulations at the investigational sites.

The Monitoring Plan is built according to a risk-based monitoring approach and describes the level of source data verification to be performed by the monitors.

Risk-based monitoring approach uses all available means to supervise the trial (central monitoring, remote monitoring and on-site monitoring), focusing in critical data points and issues ensuring that adequate monitoring (central, remote and on-site) at each site is completed to ensure protection of the rights and safety of the subjects and the quality and integrity of the data collected and submitted.

The sponsor shall provide training and the necessary guidelines to assist each investigational site on the data collection in the eCRF. Each site is responsible to report the available data requested by the CIP. In order to ensure data quality and avoid missing information in the eCRF, edit checks are designed during database development. In addition, Sponsor's CRA and Data Management team will be responsible to review the data and raise queries accordingly into the eCRF. An audit trail logging all data entered and edited is available within the EDC system. All source documents are maintained in the hospital files ready for inspection by the Sponsor and regulatory authorities upon request. The Sponsor will inform the investigator of the time period for retaining these records as per applicable regulatory requirements.

The following analysis sets will be considered for the statistical analysis :

As Treated Population This population includes all patients who were treated and undergo the studied procedure. Patients will be assigned to the study treatement groups according to the actual received treatement.

Intention-To-Treat Population This population includes all patients who have been randomized to a treatement. Patients will be assigned to the study treatement groups according to the treatement to which they have been randomized.

Per-Protocol Population This population includes all patients who were treated and undergo the studied procedure, excluding all patients with major violations to the protocol (e.g. wrong inclusion, missing data, mis-randomization, crossover, drop off before discharge). Patients will be assigned to the study treatement groups according to the treatement to which they have been randomized. All the protocol deviations will be reported in statistical report.

Assuming a rate of forearm RAO of 1% in DTRA and 3.5% in CTRA based on on two-sided alpha = 0.050 and power = 80%, 1:1 randomization needs 551 patients for each group to detect statistically significant differences in forearm RAO proportions. Then, given the crossover rate of 10% and the drop out rate of 5% for both group, at least 648 patients needs for each group to maintain proper statistical power. In total 1300 subjects will be randomized.

The primary endpoint analysis will be performed on ITT (Intention-To-Treat) population, by using two-sided superiority test with alpha = 0.05. Due to the short observation period (3 days ±2), a low number of missing data is expected. However, in case it exceeds 15-20%, missing, unused or spurious data will be considered using a tipping point analysis for each population. The comparaison in RAO rates between treatment groups will be tested by Chi-squared tests or Fisher's exact test, as appropriate. Odd-Ratio with IC95% will be calculated. Logistic regression analyses will be used to test the tendency.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient has provided written informed consent.
* Patient is undergoing diagnostic coronary angiography and/or PCI.
* Patient is willing to comply with all protocol-required evaluations during the hospitalization.
* Patient is suitable for both DTRA and CTRA using 6Fr GSS.

Exclusion Criteria:

* Patient has a medical condition that may cause non-compliance with the protocol and/or confound the data interpretation.
* Patients on chronic hemodialysis.
* Patients presenting with ST-elevated myocardial infarction (STEMI).
* Patients have chronic total occlusion (CTO) lesions in coronary artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1309 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Forearm radial artery occlusion (RAO) rate before discharge | up to 5 days
  Forearm radial artery occlusion (RAO) rate before discharge measured with Doopler Ultrasound

SECONDARY OUTCOMES:
Rate of successful sheath insertion | up to 2 days
  Rate of successful sheath insertion obtained though eCRF question
Rate of access site crossover | up to 2 days
  Rate of access site crossover - if the initial access point fails physician can perform the procedure using other access site of his/her choice This data point is captured on the eCRF
Total procedural time | up to 2 days
  Total procedural time defined as the time between initiation of local anesthesia to sheath removal - information captured on the eCRF
Sheath insertion time | up to 2 days
  Sheath insertion time recorded in the eCRF and defined as when puncture with the introducer needle first attempted until the time when introducer sheath is successfully inserted
Puncture site bleeding according to EASY criteria | up to 5 days
  Puncture site bleeding according to EASY criteria
Overall bleeding according to BARC criteria | up to 5 days
  Overall bleeding according to BARC criteria
Vascular access-site complication | up to 5 days
  Vascular access-site complication documented on the eCRF. It is composed by the rate of vessel perforation after occlusion requiring intervention, arterial dissection, pseudoaneurysm, and local haematoma
Rate of radial artery spasm | up to 2 days
  Rate of radial artery spasm captured in the eCRF. Radial arety spasm is defined as an inability to manipulate the guidewire or catheter in a smooth and pain-free manner and also as an inability to remove the sheath in a similar way at the end of the procedure
Rate of distal radial artery occlusion (dRAO) | up to 5 days
  Rate of distal radial artery occlusion (dRAO) by doopler ultrasound and capture in the eCRF
Patent hemostasis was achieved or not (CTRA) by reverse barbeau test | up to 5 days
  Patent hemostasis was achieved or not (CTRA) by reverse barbeau test
Time required to reach hemostasis | up to 5 days
  Time required to reach hemostasis, captured on the eCRF and defined as the time between sheath removal to complete hemostasis
Pain associated with the procedure: Visual Assessment Scale (VAS) | up to 5 days
  Pain associated with the procedure measured by the Visual Assessment Scale (VAS), a numeric rating scale. VAS is a 10 cm line with anchor statements on the left (no pain = 0) and on the right (worst possible pain = 10)

CONTACTS AND LOCATIONS:
Overall Officials: Adel Aminian, Dr., Principal Investigator — Hôpital Civil Marie Curie
Locations (16):
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussels Capital
  - Hôpital Civil Marie Curie, Charleroi, Hainaut
  - CHU Jolimont, Haine-Saint-Paul, Hainaut
  - UZ Brussel, Brussels
- Plzen Medical University, Pilsen, Czechia
- University Hospital Johannes Wesling Klinikum Minden, Minden, Germany
- Bács-Kiskun Megyei Kórház, Kecskemét, Hungary
- Italy (2):
  - Sant'Eugenio Hospital, Roma
  - Istituto Clinico Humanitas, Rozzano
- Shonan Kamakura General Hospital, Kanagawa, Japan
- Isala Hospital, Zwolle, Netherlands
- University Clinic of Cardiology, Skopje, Skopje, North Macedonia
- Switzerland (2):
  - HUG Geneva, Geneva
  - Kantonsspital Baselland Liestal, Liestal
- United Kingdom (2):
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiemeneij F. Left distal transradial access in the anatomical snuffbox for coronary angiography (ldTRA) and interventions (ldTRI). EuroIntervention. 2017 Sep 20;13(7):851-857. doi: 10.4244/EIJ-D-17-00079. PMID 28506941
- [Background] Corcos T. Distal radial access for coronary angiography and percutaneous coronary intervention: A state-of-the-art review. Catheter Cardiovasc Interv. 2019 Mar 1;93(4):639-644. doi: 10.1002/ccd.28016. Epub 2018 Dec 11. PMID 30536709
- [Background] Sgueglia GA, Di Giorgio A, Gaspardone A, Babunashvili A. Anatomic Basis and Physiological Rationale of Distal Radial Artery Access for Percutaneous Coronary and Endovascular Procedures. JACC Cardiovasc Interv. 2018 Oct 22;11(20):2113-2119. doi: 10.1016/j.jcin.2018.04.045. PMID 30336816
- [Background] Aminian A, Saito S, Takahashi A, Bernat I, Jobe RL, Kajiya T, Gilchrist IC, Louvard Y, Kiemeneij F, Van Royen N, Yamazaki S, Matsukage T, Rao SV. Comparison of a new slender 6 Fr sheath with a standard 5 Fr sheath for transradial coronary angiography and intervention: RAP and BEAT (Radial Artery Patency and Bleeding, Efficacy, Adverse evenT), a randomised multicentre trial. EuroIntervention. 2017 Aug 4;13(5):e549-e556. doi: 10.4244/EIJ-D-16-00816. PMID 28218605